CLINICAL TRIAL: NCT05847686
Title: A Phase 1/2 Study of a Group Model of Psilocybin-Assisted Therapy for Cancer-Related Anxiety in Patients With Metastatic Cancer
Brief Title: Psilocybin-Assisted Therapy for the Treatment of Cancer-Related Anxiety in Patients With Metastatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Principal Investigator, Anthony Back MD, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1123316; NCI-2023-02948 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020001 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-04-26; First posted 2023-05-08 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Counseling; Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (psilocybin, therapy) (Experimental): Patients receive psilocybin PO and participate in group and individual therapy sessions on trial.
  Interventions: Other: Counseling; Drug: Psilocybin; Other: Questionnaire Administration

INTERVENTIONS:
Other: Counseling — Participate in therapy visits
  Other Names: Counseling Intervention
Drug: Psilocybin — Given PO
  Other Names: CY-39; Indocybin; psilocybine
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I/II trial tests the safety and side effects of psilocybin in combination with therapy for the treatment of patients with metastatic cancer and symptoms of anxiety and/or depression. Psilocybin is a substance being studied in conjunction with therapy for the treatment of anxiety and depression in patients with cancer. In this study, the psilocybin being used is derived from the mushroom psilocybe cubensis using a patented process that results in a pharmaceutical grade version of psilocybin. Psilocybin acts by activating serotonin receptors on brain cells which can change perceptions and patterns of thinking in ways that may decrease anxiety.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive psilocybin orally (PO) and participate in group and individual therapy sessions on trial.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of metastatic solid tumor, or incurable hematologic malignancy that has been accepted by a physician in a medical record
* Measurable disease is not required
* Previous treatment with chemotherapy: There are no minimum or maximum prior lines of chemotherapy
* 18-85 years of age
* Required performance status, including the appropriate scale. Eastern Cooperative Oncology Group (ECOG) 0-2
* Hematocrit > 20
* Platelets (Plt) > 20K
* Liver function tests 1.5 x normal
* Creatinine 1.5 x normal
* Subjects of childbearing potential must be willing to use an effective contraceptive method from study enrollment until at least 1 month after receiving the investigational agent(s)
* Must be at least 4 weeks after surgery or radiotherapy at study entry, but can be receiving oral or iv chemotherapy if those schedules can be adjusted around the medication session date
* Motivated to participate in a group study and able in the research team's judgment to participate in the small group effectively
* On pre-enrollment screening tests, they will have clinically significant anxiety or depressive symptoms as defined by a score of 11 or greater on the Hospital Anxiety and Depression Scale (HADS)-Total
* English speaking- able to understand the process of consent and the risk and benefits associated with the study, and able to give written informed consent. This is a pilot study, and if future larger studies are designed, consideration will be given for non-English-speaking subjects
* Must be willing to sign a medical release for the investigators to communicate directly with their treating clinicians (mental health professional or oncologist) and doctors to confirm a medication and/or medical history
* Must provide at least one adult who is in contact with the participant at least once a day when the participant is at home who is able to verbally monitor participant-reported changes in the behavior and able to notify research staff of behavior changes that may require research staff assessment
* Has been off selective serotonin inhibitors for five half-lives of the drug plus 2 weeks
* Must avoid taking any psychiatric medications or starting a new psychiatric medication during the study. Should participant's doctor recommend starting a new psychiatric medication, participant will be required to notify the study team and the subject would withdraw from the study. (Use of prn benzodiazepines is allowed but high dose chronic benzodiazepine use must be reviewed by the principal investigator [PI]. Use of as needed [prn] gabapentoids is allowed by high dose chronic gabapentoid use must be reviewed by the PI)
* Must provide a contact (relative, spouse, close friend, or other caregiver; can be the same person) who is willing and able to be reached by the research team in the event that the participant becomes suicidal
* If the potential participant is of childbearing potential, they must have a negative pregnancy test at baseline and prior to the medication dosing session, and must agree to use adequate birth control
* Are willing to commit to preparation sessions, medication dosing sessions, integration sessions, to complete evaluation instruments and commit to be contacted for all necessary telephone contacts

Exclusion Criteria:

* Brain metastases that have not been treated
* Uncontrolled or concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy, breastfeeding, or expecting to conceive or father children for the duration of the trial through 30 days after receipt of investigational agent(s)
* Personal or immediate family history of schizophrenia, bipolar affective disorder, delusion disorder, paranoid disorder, or schizoaffective disorder
* Suicidal ideation with a Columbia-Suicidality Severity Rating Scale (C-SSRS) >= 3
* Current substance abuse disorder (although prospective subjects will not be excluded for reasonable alcohol use that does not meet criteria for alcohol use disorder or marijuana use that does not meet criteria for substance use disorder)
* Neuroleptic (including olanzapine, prochlorperazine, promethazine), and selective serotonin reuptake inhibitor (SSRI) medications that cannot be tapered and discontinued in conjunction with the participant's prescribing physician (although ondansetron can be used for nausea)
* Unstable neurological or medical condition; history of seizure, chronic/severe headaches
* Any use of psychedelic drugs in high doses (psilocybin > 2 grams of dried mushrooms, LSD > 200 micrograms) within the prior 12 months (microdosing will not require exclusion but participants would have to agree to discontinue microdosing 1 month before study entry)
* Use of tramadol, due to the potential for serotonin syndrome with concomitant use of psilocybin
* Individuals who are on MOAI (monoamine oxidase inhibitors) or who have a known sensitivity to the drug or its metabolites. Psilocybin is contraindicated in medications that are known UGT (UDP-glucuronosyltransferase) enzyme modulators. The concurrent use of SSRI/serotonin-norepinephrine reuptake inhibitor (SNRI) meds is assumed to be contraindicated due to the potential to increase the risk of serotonin syndrome and/or to attenuate the binding of psilocin to the HT2A receptor
* A marked baseline prolongation of QT/corrected QT (QTc) interval (e.g., demonstration on > 1 electrocardiogram (ECG) of a QTc interval > 450 milliseconds (ms)
* A history of additional risk factors for Torsade de Points (including but not limited to: heart failure, hypokalemia, family history of long QT syndrome)
* The use of concomitant medications that prolong the QT/QTc interval

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Back, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Back A, Myers S, Guy J, Perez J, Lazar Thorn L, McGregor B. Evolving Guidelines for the Use of Touch During a Clinical Trial of Group Psilocybin-Assisted Therapy. Psychedelic Med (New Rochelle). 2024 Dec 2;2(4):187-191. doi: 10.1089/psymed.2023.0069. eCollection 2024 Dec. PMID 40051480

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Psilocybin, Therapy)
Started | 55
Completed | 52
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Psilocybin, Therapy)
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 53 [26 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 49
  More than one race | 1
  Unknown or Not Reported | 0
Hospital Anxiety and Depression Scale [Mean (Standard Deviation); unit: units on a scale] | 17.5 (5.99)

OUTCOME MEASURES:

1. Primary Outcome: Number of Instances of Potentially Unattended Psilocybin-related Distress During Psilocybin Sessions.
Description: Defined as the occurrence of participant distress among study participants in the small group during the psilocybin administration session on Day 0 that requires 1:1 facilitator attention that cannot be met by the 4-person facilitation team. The size of small groups of different sizes will vary over the course of the study. Descriptive statistics will be used to analyze and will be tabulated on Day 0 after each group intervention. Backup facilitators will be available when this occurs.
Time Frame: At psilocybin administration session on day 0
Measure: Number; unit: Events
Arm/Group | Treatment (Psilocybin, Therapy)
Number analyzed (Participants) | 52
Events | 0

2. Secondary Outcome: Change in Measured Anxiety and Depression: Hospital Anxiety and Depression Scale (HADS)
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-administered measure of depression and anxiety. The HADS is not a diagnostic tool, but can screen for anxiety and depression. The HADS has 14 items in total and asks about mood in the past week. Seven items assess depression and seven items assess anxiety. The HADS can be administered repeatedly without impacting on validity. Each item is rated on a 4-point scale and the total provides a score of 0 minimum up to 21 maximum. A higher score indicates higher distress.
Time Frame: From 14 days before the psilocybin session to 28 days (4 weeks) after the psilocybin session
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment (Psilocybin, Therapy)
Number analyzed (Participants) | 52
units on a scale | -7.29 [-9.33 to -5.25]
Statistical Analysis 1: Comparison: Treatment (Psilocybin, Therapy); Test type: Other; p < .0001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment (Psilocybin, Therapy)
All-Cause Mortality (participants affected / at risk) | 2/52
Serious Adverse Events (participants affected / at risk) | 3/52
Other Adverse Events (participants affected / at risk) | 30/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Psilocybin, Therapy) (N=52)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — Death from progressive cancer
dehydration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — chemotherapy-related dehydration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Psilocybin, Therapy) (N=52)
hypertension (Cardiac disorders) | 19 (19) — psilocybin-related hypertension
anxiety (Nervous system disorders) | 3 (3) — psilocybin-related anxeity
headache (Nervous system disorders) | 2 (2) — mild
nausea (Gastrointestinal disorders) | 2 (2) — psilocybin-related nausea
shaking (Musculoskeletal and connective tissue disorders) | 1 (1) — psilocybin-related somatic reaction
malaise (Psychiatric disorders) | 2 (2) — immediately after psilocybin
chest tightness, muscular (Musculoskeletal and connective tissue disorders) | 1 (1)
migraine (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a single arm open label Phase 1-2 study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT05847686/Prot_SAP_002.pdf
  • Informed Consent Form (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT05847686/ICF_000.pdf